CLINICAL TRIAL: NCT04604587
Title: MRI-visible Enlarged Perivascular Spaces and the Alteration of Lymphatic Drainage System in Cerebral Amyloid Angiopathy
Brief Title: MRI-visible Enlarged Perivascular Spaces and the Alteration of Lymphatic Drainage System in CAA
Acronym: CAA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201912003MINC
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Cerebral Amyloid Angiopathy; Intracerebral Hemorrhage
Keywords: Cerebral Amyloid Angiopathy; Intracerebral Hemorrhage; Magnetic resonance imaging; Position emitting topography
MeSH Terms: conditions — Cerebral Amyloid Angiopathy; Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- amyloid PET、T807 PET (Experimental): PET/CT
  Interventions: Drug: 1. amyloid PET；2. T807 PET

INTERVENTIONS:
Drug: 1. amyloid PET；2. T807 PET — 1. Dynamic PET acquisition for 70 minutes will be acquired after injection of 10±5 mCi 11C-PiB
  2. Dynamic PET imaging 3D acquisition will be acquired 80 minutes after injection of 10 mCi 18F-T807

SUMMARY:
In this three-year proposal, we will explore the MRI-visible EPVS in CAA and investigate its pathophysiology using animal models. Our specific aims include: (1) Establish the relationship of MRI-visible enlarged perivascular space and CAA, (2) Determine whether vascular amyloid clearance in CAA is associated with lymphatic drainage system, (3) Establish longitudinal data for MRI-visible enlarged perivascular space and cerebral amyloid angiopathy progression.

DETAILED DESCRIPTION:
Cerebral amyloid angiopathy (CAA) involves amyloid deposition in the vessel walls in the cerebral cortex and overlying leptomeninges, causing symptomatic intracerebral lobar intracerebral hemorrhage (ICH) in the elderly. CAA is considered as a form of cerebral small vessel disease, which refers to a group of vascular pathologies that affect the small vessels of the brain. In addition to lobar ICH, patients may present with other parenchymal injuries that can be detected on blood-sensitive MRI, such as multiple strictly lobar cerebral microbleeds, cortical superficial siderosis and leukoariosis. Recently, CAA has been suggested in association with MRI-visible enlarged perivascular space (EPVS) in centrum-semiovale (CSO), contrary to more severe MRI-visible EPVS in basal ganglia that is frequently found in chronic hypertension. The dilated perivascular space in CAA is suggestive of chronic poor perivascular drainage of the leptomeningeal arteries, predisposing individuals to impaired or altered meningeal lymphatic drainage and causing defect in amyloid clearance and subsequent CAA development. Nevertheless, it is unknown whether lymphatic drainage are the main routes for vascular amyloid clearance, and its relationship to the long-term outcome has not been clearly investigated in clinical patients yet.

In this three-year proposal, we will explore the MRI-visible EPVS in CAA and investigate its pathophysiology using animal models. Our specific aims include: (1) Establish the relationship of MRI-visible enlarged perivascular space and CAA, (2) Determine whether vascular amyloid clearance in CAA is associated with lymphatic drainage system, (3) Establish longitudinal data for MRI-visible enlarged perivascular space and cerebral amyloid angiopathy progression. In the first year, we will recruit spontaneous ICH patients for brain MRI, in vivo amyloid imaging and measuring their plasma Aβ40/42 levels. We aim to confirm EPVS in CSO as a specific marker for CAA, and to provide direct evidence that dilated perivascular space is worse with more advanced CAA; For the second year, we plan to use transgenic CAA mouse models to confirm that meningeal lymphatic drainage routes are crucial for clearance of vascular amyloid-β. We will manipulate the lymphatic drainage routes by either blockage or enhancement of the lymphatic vessels, to see if the vascular amyloid clearance is affected; For the third year, the main research focus will on be establishing the longitudinal data on amyloid and tau deposition in clinical ICH patients. We plan to repeat in vivo amyloid imaging in 2 years, for the purpose of validating our hypothesis in human that baseline worse lymphatic drainage function is associated with quicker cerebral vascular amyloid progression or prediction of future CAA development. We will also recruit patients for in vivo tau imaging to investigate long-term neuronal injury and neurodegeneration, namely tau-mediated neurofibrillary tangle, in relation to the impaired perivascular drainage in CAA.

ELIGIBILITY:
Inclusion Criteria:

1. Age：above 20 years old.
2. Evidence of intraparenchymal hemorrhage on CT or MRI.
3. Patient agrees to participate in the study and receive neurophsychological examinations, genetic and biochemical markers test, MRI and PET imaging.

Exclusion Criteria:

1. patients with potential causes of hemorrhage including trauma, structural lesion, brain tumor, or coagulopathy due to systemic disease or medication.
2. Patients could not receive the PET and MRI studies, including but not limited to poor cooperative agitation impeding adequate study, allergy to contrast medium, hemodynamic instability, implantation of cardiac pacemaker, past history of receiving aneurysm clipping, panic mood to MRI study, impaired kidney function.
3. Patients with pregnancy or recently having a plan for pregnancy.
4. Patients with breast feeding or recently having a plan for breast feeding.
5. Patients with history of allergy to 11C-PiB and 18F-T807, or severe allergy history.
6. Patient or family who does not agree to participate in the study.
7. patient with high risk by doctor evaluate.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
PET imaging | in 3 days
  PET data will reconstruct with ordered set expectation maximization, corrected for attenuation, and each frame will be evaluated to verify adequate count statistics and absence of head motion.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No